CLINICAL TRIAL: NCT00083122
Title: Phase II Trial of Flavopiridol and Cisplatin in Advanced Epithelial Ovarian and Primary Peritoneal Carcinomas
Brief Title: Cisplatin and Flavopiridol in Treating Patients With Advanced Ovarian Epithelial Cancer or Primary Peritoneal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2009-00029; NCI-2009-00029 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000363562; MC0261 (Other: Mayo Clinic); 5876 (Other: CTEP); N01CM62205 (NIH); P30CA015083 (NIH)
Record Dates: First submitted 2004-05-14; First posted 2004-05-17 (Estimated); Results first posted 2013-05-14 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2013-04

CONDITIONS: Recurrent Ovarian Epithelial Cancer; Recurrent Primary Peritoneal Cavity Cancer; Stage IIIA Ovarian Epithelial Cancer; Stage IIIA Primary Peritoneal Cavity Cancer; Stage IIIB Ovarian Epithelial Cancer; Stage IIIB Primary Peritoneal Cavity Cancer; Stage IIIC Ovarian Epithelial Cancer; Stage IIIC Primary Peritoneal Cavity Cancer; Stage IV Ovarian Epithelial Cancer; Stage IV Primary Peritoneal Cavity Cancer
MeSH Terms: conditions — Carcinoma, Ovarian Epithelial | interventions — Cisplatin; alvocidib

ARMS (2):
- Group 1 (Experimental): Patients receive cisplatin IV over 30 minutes and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: alvocidib; Drug: cisplatin/flavopiridol
- Group 2 (Experimental): Patients receive cisplatin IV over 30 minutes and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: cisplatin; Drug: alvocidib; Drug: cisplatin/flavopiridol

INTERVENTIONS:
Drug: cisplatin — Given IV
  Other Names: CACP; CDDP; CPDD; DDP
Drug: alvocidib — Given IV
  Other Names: FLAVO; flavopiridol; HMR 1275; L-868275
Drug: cisplatin/flavopiridol — Given IV

SUMMARY:
This phase II trial is studying how well giving cisplatin together with flavopiridol works in treating patients with advanced ovarian epithelial cancer or primary peritoneal cancer. Drugs used in chemotherapy, such as cisplatin and flavopiridol, work in different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

DETAILED DESCRIPTION:
OBJECTIVES:

I. Determine the response rate, time to progression, and survival in patients with advanced ovarian epithelial or primary peritoneal cancer treated with cisplatin and flavopiridol.

II. Determine the toxicity of this regimen in these patients.

OUTLINE: This is a multicenter study. Patients are accrued to two separate groups (Group 2 closed to accrual as of 3/10/06) .

GROUP 1: Patients receive cisplatin IV over 30 minutes and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

GROUP 2 (Closed to accrual as of 3/10/06): Patients receive cisplatin IV over 30 minutes and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months for up to 3 years.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed ovarian epithelial or primary peritoneal cancer:

Advanced disease

* Meets at least 1 of the following criteria:

  * Measurable disease;
  * Evaluable disease plus CA 125 >= 2 times post-treatment nadir
* Treated with 1, and only 1, prior platin-containing chemotherapy regimen (e.g., paclitaxel or carboplatin-based) for ovarian epithelial or primary peritoneal cancer
* Prior treatment with the same regimen at first relapse allowed;

  * No more than 3 total chemotherapy regimens allowed provided exactly 1 has been platin-containing;
  * Must also have platin-resistant disease as defined for Group 1;
  * Rechallenge with a single regimen upon progression after a hiatus from therapy counts as a single regimen
* Group 1, meeting 1 of the following criteria:

  * Patients who relapse during or < 6 months after completion of post-debulking chemotherapy;
  * "Platinum sensitive" patients in second relapse after having been treated/rechallenged with their initial regimen upon first relapse
* Group 2 (Closed to accrual as of 3/10/06):

  * Patients who relapse >= 6 months after completion of post-debulking chemotherapy and are not retreated with the same or a different regimen
* No CNS metastases
* Performance status:

  * ECOG 0-2
* Hematopoietic:

  * Absolute neutrophil count >= 1,500/mm3;
  * Platelet count >= 100,000/mm3;
  * Hemoglobin >= 10 g/dL (Note: May be supported with transfusion, epoetin alfa, or darbepoetin alfa)
* Hepatic:

  * AST =< 2.5 times upper limit of normal (ULN);
  * Alkaline phosphatase =< 2.5 times ULN;
  * Bilirubin =< 1.5 times ULN
* Renal:

  * Creatinine =< 1.5 times ULN
* Cardiovascular:

  * No cardiac arrhythmia;
  * No cardiac failure
* Not pregnant or nursing
* Negative pregnancy test
* More than 3 weeks since prior chemotherapy (6 weeks for nitrosoureas)
* More than 3 weeks since prior radiotherapy
* Recovered from all prior therapy
* Fertile patients must use effective contraception
* No other malignancy within the past 5 years except non-melanoma skin cancer or carcinoma in situ of the cervix
* No diabetes
* No peripheral neuropathy >= grade 2
* No baseline diarrhea (>= 4 stools/day)
* No uncontrolled infection
* No other concurrent uncontrolled serious medical condition
* No concurrent routine colony-stimulating factors

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2004-04; Primary Completion 2010-07 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Keith Bible, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

REFERENCES:
- [Derived] Bible KC, Peethambaram PP, Oberg AL, Maples W, Groteluschen DL, Boente M, Burton JK, Gomez Dahl LC, Tibodeau JD, Isham CR, Maguire JL, Shridhar V, Kukla AK, Voll KJ, Mauer MJ, Colevas AD, Wright J, Doyle LA, Erlichman C; Mayo Phase 2 Consortium (P2C); North Central Cancer Treatment Group (NCCTG). A phase 2 trial of flavopiridol (Alvocidib) and cisplatin in platin-resistant ovarian and primary peritoneal carcinoma: MC0261. Gynecol Oncol. 2012 Oct;127(1):55-62. doi: 10.1016/j.ygyno.2012.05.030. Epub 2012 Jun 1. PMID 22664059

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Forty-five patients were enrolled between December 23, 2004 and February 25, 2010: 40 patients to Group 1 (platin resistant; 14 evaluable, 26 measurable) and 5 patients to Group 2 (platin sensitive; 1 evaluable, 4 measurable). Group 2 was closed on 03/10/2006 due to poor accrual.
Pre-assignment Details: Participants who progressed or relapsed during or within 6 months of primary platinum-based therapy constituted Group 1 ("Platin Resistant"). Participants who relapsed > 6 months following completion of platinum-based therapy, and who had received only a single prior chemotherapy regimen constituted Group 2 ("Platin Sensitive").
Groups:
- Group 1 (Platin Resistant); Group 2 (Platin Sensitive): Patients receive 60 mg/m^2 of cisplatin IV over 2 hours and 100 mg/m^2 flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Period: Overall Study
Arm/Group | Group 1 (Platin Resistant) | Group 2 (Platin Sensitive)
Started | 40 | 5
Completed | 40 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Group 1 (Platin Resistant); Group 2 (Platin Sensitive): Patients receive cisplatin IV over 2 hours and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
- Total: Total of all reporting groups
Arm/Group | Group 1 (Platin Resistant) | Group 2 (Platin Sensitive) | Total
Number analyzed (Participants) | 40 | 5 | 45
Age, Continuous [Median (Full Range); unit: years] | 59 [29 to 79] | 61 [41 to 73] | 59 [29 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 5 | 45
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 40 | 5 | 45

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Confirmed Tumor Responses Defined to be Either a Complete Response (CR) or Partial Response (PR)
Description: A Complete Response (CR) is defined as the disappearance of all target lesions and normalization of tumor biomarkers.
  A Partial Response (PR) is defined as at least a 30% decrease in the sum of the LD of target lesions taking as reference the baseline sum LD.
  A confirmed tumor response is defined to be either a CR or PR noted as the objective status on 2 consecutive evaluations at least 4-6 weeks apart.
Time Frame: 24 weeks
Population: All 45 participants were analyzed.
Measure: Number; unit: Percentage of Participants
Groups:
- Group 1 (Platin Resistant); Group 2 (Platin Sensitive): Patients receive 60 mg/m^2 cisplatin IV over 2 hours and 100 mg/m^2 flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group 1 (Platin Resistant) | Group 2 (Platin Sensitive)
Number analyzed (Participants) | 40 | 5
Percentage of Participants
  Complete Response (CR) | 2.5 | 0
  Partial Response (PR) | 15 | 40

2. Secondary Outcome: Overall Survival
Description: Will be estimated using the method of Kaplan-Meier.
Time Frame: Time from registration to date of last follow-up or death due to any cause, assessed up to 3 years
Population: All 40 participants in Group 1 were analyzed for this primary endpoint. However, due to the low accrual and early group 2 closure, Group 2 was not statistically evaluated for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Group 2 (Platin Sensitive): Patients receive 60 mg/m^2cisplatin IV over 2 hours and 100 mg/m^2 flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group 1 (Platin Resistant) | Group 2 (Platin Sensitive)
Number analyzed (Participants) | 40 | 0
months | 17.5 [10.8 to 24.5] |

3. Secondary Outcome: Time to Progression
Description: Time to progression will be estimated using the method of Kaplan-Meier. Progression is defined as having at least a 20% increase in the sum of longest diameter (LD) of target lesions taking as reference the smallest sum LD recorded since the treatment started or the appearance of one or more new lesions.
Time Frame: Time from registration to the date of progression or last follow-up, assessed up to 3 years
Population: All 40 participants from Group 1 were analyzed. However, due to slow accrual and early closure, Group 2 was not statistically analyzed for this endpoint.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Group 1 (Platin Resistant) | Group 2 (Platin Sensitive)
Number analyzed (Participants) | 40 | 0
months | 4.3 [2.89 to 5.81] |

ADVERSE EVENTS:
Groups:
- Group 1 and Group 2 Combined: Patients receive cisplatin IV over 2 hours and flavopiridol IV over 24 hours on day 1. Courses repeat every 3 weeks in the absence of disease progression or unacceptable toxicity.
Arm/Group | Group 1 and Group 2 Combined
Serious Adverse Events (participants affected / at risk) | 23/45
Other Adverse Events (participants affected / at risk) | 45/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 and Group 2 Combined (N=45)
Arrhythmia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1)
Hearing impaired (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 2 (2)
Diarrhea (Gastrointestinal disorders) | 1 (1)
Nausea (Gastrointestinal disorders) | 4 (4)
Small intestinal obstruction (Gastrointestinal disorders) | 3 (3)
Vomiting (Gastrointestinal disorders) | 3 (3)
Chest pain (General disorders) | 1 (1)
Fatigue (General disorders) | 2 (2)
Fever (General disorders) | 2 (3)
Gallbladder obstruction (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 3 (3)
Pneumonia (Infections and infestations) | 1 (1)
Creatinine increased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 4 (4)
Serum magnesium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 1 (1)
Serum potassium decreased (Metabolism and nutrition disorders) | 2 (2)
Serum sodium decreased (Metabolism and nutrition disorders) | 1 (1)
Ataxia (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 2 (2)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pruritus (Skin and subcutaneous tissue disorders) | 1 (1)
Skin disorder (Skin and subcutaneous tissue disorders) | 1 (1)
Sweating (Skin and subcutaneous tissue disorders) | 1 (1)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 and Group 2 Combined (N=45)
Hemoglobin decreased (Blood and lymphatic system disorders) | 42 (179)
Palpitations (Cardiac disorders) | 2 (2)
Hearing impaired (Ear and labyrinth disorders) | 2 (3)
Hearing test abnormal (Ear and labyrinth disorders) | 1 (1)
Tinnitus (Ear and labyrinth disorders) | 3 (15)
Abdominal pain (Gastrointestinal disorders) | 1 (1)
Colitis (Gastrointestinal disorders) | 1 (1)
Constipation (Gastrointestinal disorders) | 3 (7)
Diarrhea (Gastrointestinal disorders) | 31 (123)
Dry mouth (Gastrointestinal disorders) | 1 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (4)
Ear, nose and throat examination abnormal (Gastrointestinal disorders) | 1 (1)
Gastritis (Gastrointestinal disorders) | 1 (5)
Mucositis oral (Gastrointestinal disorders) | 5 (5)
Nausea (Gastrointestinal disorders) | 42 (153)
Vomiting (Gastrointestinal disorders) | 32 (93)
Fatigue (General disorders) | 44 (165)
Pain (General disorders) | 2 (7)
Urinary tract infection (Infections and infestations) | 1 (1)
Vascular access complication (Injury, poisoning and procedural complications) | 1 (1)
Alanine aminotransferase increased (Investigations) | 1 (1)
Alkaline phosphatase increased (Investigations) | 15 (37)
Aspartate aminotransferase increased (Investigations) | 9 (15)
Blood bilirubin increased (Investigations) | 1 (1)
Creatinine increased (Investigations) | 12 (29)
Leukocyte count decreased (Investigations) | 14 (30)
Neutrophil count decreased (Investigations) | 33 (59)
Platelet count decreased (Investigations) | 28 (90)
Weight loss (Investigations) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 12 (18)
Blood glucose increased (Metabolism and nutrition disorders) | 32 (74)
Blood uric acid increased (Metabolism and nutrition disorders) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 2 (2)
Serum albumin decreased (Metabolism and nutrition disorders) | 7 (11)
Serum calcium decreased (Metabolism and nutrition disorders) | 6 (9)
Serum calcium increased (Metabolism and nutrition disorders) | 1 (2)
Serum magnesium decreased (Metabolism and nutrition disorders) | 24 (77)
Serum magnesium increased (Metabolism and nutrition disorders) | 2 (2)
Serum phosphate decreased (Metabolism and nutrition disorders) | 2 (2)
Serum potassium decreased (Metabolism and nutrition disorders) | 11 (13)
Serum potassium increased (Metabolism and nutrition disorders) | 1 (1)
Serum sodium decreased (Metabolism and nutrition disorders) | 10 (21)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Myalgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Tumor pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Dysgeusia (Nervous system disorders) | 2 (5)
Extrapyramidal disorder (Nervous system disorders) | 1 (2)
Headache (Nervous system disorders) | 3 (4)
Peripheral motor neuropathy (Nervous system disorders) | 3 (10)
Peripheral sensory neuropathy (Nervous system disorders) | 33 (114)
Anxiety (Psychiatric disorders) | 1 (1)
Cough (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 (6)
Alopecia (Skin and subcutaneous tissue disorders) | 9 (11)
Body odor (Skin and subcutaneous tissue disorders) | 1 (1)
Rash acneiform (Skin and subcutaneous tissue disorders) | 2 (8)
Hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 4 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less